CLINICAL TRIAL: NCT03896178
Title: Early Detection of Prostate Cancer in Firefighters - a Register-based Study of Prognostic Factors and Survival
Brief Title: Prostate Cancer in Firemen: Early Diagnosis Because of Increased Diagnostic Pressure?
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Institute of Public Health (Other Government); Extrastiftelsen (Other); The National Institute of Occupational Health (Unknown); Norwegian Confederation of Trade Unions (Unknown); Fagforbundet (Unknown); Gjensidige Foundation (Unknown); Norwegian Cancer Society (Other); Norwegian Firefighters Fight Cancer (Unknown); Norwegian Labour Inspection Authority (Unknown)
Responsible Party: Principal Investigator, Jarle Jakobsen, PhD-student, Norwegian Institute of Public Health
Other Study IDs: 2019/542
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 60 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Firefighters
  Interventions: Other: None, observational study
- Pilots
  Interventions: Other: None, observational study
- Police
  Interventions: Other: None, observational study
- Military personnel
  Interventions: Other: None, observational study
- Controls: Control group matched for geographic location (county), and year of diagnosis. Consisting of all other workers than the four specified groups.
  Interventions: Other: None, observational study

INTERVENTIONS:
Other: None, observational study — None, observational study

SUMMARY:
Firefighters, police, military personnel and pilots are all shown to have a higher incidence of prostate cancer than the general population. A possible explanation for this is that these four groups of employees need regular mandatory health-checkups. If these checkups increase the chances of having a PSA or DRE performed one could expect the workers in question to have a higher probability than the general population of being diagnosed with prostate cancer. If this is the case the four groups should have cancers that are lower grade and have better survival. The investigators wish to examine this by comparing the four groups with a control group made up of all other workers with regards to prognostic factors at the time of diagnosis and survival rates. This will be done by extracting data from the Cancer Registry of Norway, coupled with employment data from Statistics Norway. This study is also a part of a project on cancer in firefighters. If the prostate cancers in firefighters differ significantly from the other three specified groups, this could point to an exposure specific for firefighters, e.g. fire smoke, as an etiologic factor.

ELIGIBILITY:
Inclusion Criteria:

* All cases of prostate cancer as registered by the Cancer Registry of Norway

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All men registered in the Cancer Registry of Norway with prostate cancer. Analysis of firefighters, pilots, police, military personnel and a matched group of other workers.
Sampling Method: Non-Probability Sample
Enrollment: 137536 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
Cause-specific mortality rate for prostate cancer | From January 1st 1960 until December 31st 2018

SECONDARY OUTCOMES:
TNM staging | January 1st 1960 until December 31st 2018
Gleason score | January 1st 1960 until December 31st 2018
  Score based on microscopic appearance of prostate cancer tissue. Sum of two scores, each ranging from 1-5 (only whole numbers), meaning the final score ranges from 2-10. A higher score is associated with a more aggressive/less differentiated tumor. It is normal to group scores 2-6 together in >7. It is also normal to differentiate between 7 (4+3) (worse), and 7 (3+4) (better).
PSA at time of diagnosis | January 1st 1960 until December 31st 2018
Functional status at time of diagnosis (WHO classification) | January 1st 1960 until December 31st 2018

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Registry of Norway, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No